CLINICAL TRIAL: NCT03561818
Title: Comparison of Pulmonary Rehabilitation Efficiency in Home-based With Hospital-based Pulmonary Rehabilitation in Bronchiectasis
Brief Title: Comparison of PR Efficiency in Home-based With Hospital-based PR in Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR_bronchiectasis
Record Dates: First submitted 2018-05-14; First posted 2018-06-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Bronchiectasis; Pulmonary Rehabilitation; Lung Diseases; Lung Diseases, Interstitial
MeSH Terms: conditions — Bronchiectasis; Lung Diseases; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-based group (Experimental): 2 months hospital-based pulmonary rehabilitation program
  Interventions: Other: Hospital-based pulmonary rehabilitation
- Home-based group (Experimental): 2 months home-based pulmonary rehabilitation program
  Interventions: Other: Home-based pulmonary rehabilitation

INTERVENTIONS:
Other: Hospital-based pulmonary rehabilitation — The patients who undergo two days pulmonary rehabilitation under supervision in our clinic and three days a week at home during two months will taken as hospital group. The exercises include breathing exercises, treadmill (15sc), cycle training (15sc), arm ergometer training (15sc), peripheral muscle training and stretching exercises with free weights.
  Arms: Hospital-based group
Other: Home-based pulmonary rehabilitation — The patients who follow a home-based pulmonary rehabilitation program for two months comprising breathing exercises, training in chest hygiene techniques, peripheral muscle strengthening training and self-walking for 5 days in a week for two months. An exercise follow-up form will give to the patients to record their daily exercises. A similar form will fill by physiotherapist once a week during phone call.
  Arms: Home-based group

SUMMARY:
The investigators aimed to compare the home-based Pulmonary Rehabilitation with the hospital-based pulmonary rehabilitation in terms of pulmonary rehabilitation efficiency in patient with bronchiectasis.

DETAILED DESCRIPTION:
While the benefits of pulmonary rehabilitation (PR) in cases of chronic obstructive pulmonary disease (COPD) have been well-documented, there have been only a limited number of studies investigating the efficacy of PR in patients with bronchiectasis. Some of these studies have reported positive effects of PR also in bronchiectasis patients, but have underlined the need for additional studies including larger patient groups to define PR indications, and to ensure that exercise protocols are specific for this patient group. There are many PR organizational types, such as hospital-based, telephone-mentoring with home-based or tele monitorization programs. Hospital-based supervised programs are time-consuming and costly practices. For this reason, there is a need for further studies on the effectiveness and benefits of unsupervised programs. In this study, we will compare unsupervised home-based PR and supervised hospital-based PR in terms of pulmonary rehabilitation effectiveness.

The pulmonary function tests, dyspnea perception, quality of life and exercise capacity assessments will performed before and after pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70
* Patients signing informed consent form
* Bronchiectasis patients in the stable phase who were diagnosed with High-resolution computed tomography (HRCT).

Exclusion Criteria:

* Decompensated heart failure, uncontrolled hypertension (Systolic Blood Pressure> 200, Diastolic Blood Pressure> 110),
* Additional diseases that may prevent exercise,
* To be regularly exercising regularly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline the 6-minute walking distance at two months. | Two months
Changes from baseline the modified Medical Research Council (mMRC) scale at two months. | Two months
  Dyspnea perceptions during daily life activities will assess according to the modified Medical Research Council (mMRC) scale. The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "0" means no dyspnea perception, "4" means severe dyspnea perception.

SECONDARY OUTCOMES:
Changes from baseline the forced expiratory volume in one second at two months. | Two months
  The Pulmonary Function Test conducted using a Sensor Medics model 2400 device (Yorba Linda, CA, USA), in line with American Thoracic Society (ATS) guidelines.
Changes from baseline the peripheral muscle strength at two months. | Two months
  Peripheral Muscle Strength will measure using a digital dynamometer(J-Tech Commander muscle testing device), with three measurements make in total of the quadriceps femoris, tibialis anterior and iliopsoas muscles.
Changes from baseline the Quality of Life at two months. | Two months
  St. George Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided